CLINICAL TRIAL: NCT00771446
Title: Safety & Efficacy of the Extracorporeal Liver Assist Device (ELAD) in Patients With Acute on Chronic Hepatitis (AOCH)
Brief Title: Safety & Efficacy of the Extracorporeal Liver Assist Device (ELAD) System in Patients With Hepatic Insufficiency
Acronym: ELAD
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vital Therapies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VTI-201
Record Dates: First submitted 2008-10-09; First posted 2008-10-13 (Estimated); Last update posted 2013-04-12 (Estimated); Status verified 2013-04

CONDITIONS: Acute Hepatitis; Chronic Hepatitis
Keywords: Hepatitis, acute; Acute Hepatitis OR Chronic Hepatitis
MeSH Terms: conditions — Hepatitis, Chronic; Hepatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ELAD (plus Standard of Care) (Experimental): Treatment with ELAD in addition to standard of care therapy Standard of care therapy defines uniform treatment for ascites, esophageal varices, dietary recommendations, etc.
  Interventions: Biological: ELAD plus standard of care treatment; Other: Standard of care treatment
- Standard of Care (Control) (Other): Standard of care treatment Standard of care for acute liver failure patients including medications and treatments typically given to these patients (Pentoxifylline, corticosteroids, abdominal paracentesis, nutritional therapy, etc., if indicated)
  Interventions: Other: Standard of care treatment

INTERVENTIONS:
Biological: ELAD plus standard of care treatment — ELAD is a liver assist system - Standard of care for acute liver failure patients including medications and treatments typically given to these patients (Pentoxifylline, corticosteroids, abdominal paracentesis, nutritional therapy, etc., if indicated)
  Arms: ELAD (plus Standard of Care)
Other: Standard of care treatment — Standard of care for acute liver failure patients including medications and treatments typically given to these patients (Pentoxifylline, corticosteroids, abdominal paracentesis, nutritional therapy, etc., if indicated)

SUMMARY:
Evaluate on how well the ELAD system works in treating people with liver failure.

DETAILED DESCRIPTION:
This is a multicenter, open-label, randomized, concurrent control study of subjects with acute on chronic hepatitis. Subjects meeting the eligibility requirements of the study will be randomly assigned in a 2:1 ratio to receive either standard medical therapy for acute liver failure plus the ELAD system, or standard medical therapy alone, with the latter defined as conventional therapy for acute on chronic hepatitis determined to be clinically appropriate by the treating physician.

Immediately prior to treatment initiation, subject eligibility will be confirmed. Treatment with ELAD will continue for a minimum of 3 days and up to a maximum of 10 days or until clinical status improves relative to study entry. Subjects will be followed until 30 days has elapsed since study enrollment (control) or 30 days has elapsed since cessation of ELAD therapy (ELAD group), whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

1. Weight >40 kilograms
2. Age >18 and <70 years
3. Acute decompensation of cirrhosis over the preceding 48-72 hour period
4. Up to 4 weeks from symptom onset to presentation
5. Presence of a precipitating event
6. Either a MELD score of ≥32, or ≥24 with one or more of the following

   * Severe encephalopathy of grade 3 or 4 on the Westhaven scale
   * Renal dysfunction typical of type-1 hepato-renal syndrome, i.e. acute renal failure without evidence of elevated serum creatinine (>2.5mg/dL) during the 1 to 6 months prior to study entry. Serum creatinine at study entry >2.5mg/dL does not exclude the subject from enrolment
7. SOFA score ≥9 at the initial Screening Visit

Exclusion Criteria:

1. Platelets <50,000 or reducing to <80,000 over a 72 hour period
2. Renal failure: Serum creatinine ≥2.5 mg/dL as measured during the 1 - 6 month period prior to study entry. If a subject has a contraindication to renal replacement therapy (hemodialysis or hemofiltration), then the subject should be excluded from entry into the study
3. Active sepsis. Sepsis will be defined as positive microbiological culture, ascitic white cell count >450 cells/mm³ (or ascitic neutrophil count >250 cells/mm³), or clinical signs and chest x-ray appearances for at least 48 hours without clinical improvement prior to randomization, or other evidence of infection not under control
4. Evidence of major hemorrhage indicated by requiring ≥ 4 unit blood transfusion within a 24 hour period, or hemodynamic instability (sustained pulse >120 beats/min and systolic blood pressure <100 mmHg over one hour). Subjects with a recent history of gastrointestinal hemorrhage who have been successfully treated and remain hemodynamically stable for a period of 48 hours will then be eligible for the study
5. Evidence (by physical exam, history, or laboratory evaluation) of significant concomitant disease including chronic congestive heart failure, vascular disease, emphysema, AIDS, fatty-liver disease of non-alcoholic origin, hepatitis due to herpes virus, Wilson's disease, or Budd-Chiari syndrome;
6. Known history of hepatocellular carcinoma beyond the Milan criteria and/or portal vein thrombosis
7. Evidence of Small Bowel Perforation within 48 hours of treatment;
8. Evidence of brain death as determined by blood flow studies positive for herniation and/or absence of pupillary reflex
9. Mean Arterial Pressures (MAP) < 50 mm Hg for one hour or longer;
10. Requirement for escalating doses of vasopressor support of an alpha-adrenergic agent for one hour or longer and evidence of hemodynamic instability;
11. Clinical or radiographic evidence of a new stroke or intracerebral bleeding
12. Seizures uncontrolled by medication
13. Acute myocardial infarction based on clinical and/or electrocardiographic evidence
14. Lung disease defined by a PaO2 <60 mm Hg or a history of severe COPD or interstitial lung disease
15. Pregnancy as determined by βHCG results, or lactation
16. Participation in another investigational drug, biologic, or device study within one month of enrollment

Ages: 19 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-10; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
To provide evidence that (1) subjects treated with ELAD have a higher 30-day transplant-free survival in subjects with AOCH than those not treated with ELAD, and (2) it is safe when used for 3 to 10 days of treatment. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Todd Frederick, MD, Principal Investigator — California Pacific Medical Center; Donald Hillebrand, MD, Principal Investigator — Scripps Green Hospital; Helen Te, MD, Principal Investigator — University of Chicago; Robert Brown, MD, Principal Investigator — Columbia University; Lena Napolitano, MD, Principal Investigator — University of Michigan Hospital; Winfred Williams, MD, Principal Investigator — Massachusetts General Hospital
Locations (6):
- United States (6):
  - Scripps Clinic, La Jolla, California
  - California Pacific Medical Center, San Francisco, California
  - University of Chicago Medical Center, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan Hospital, Ann Arbor, Michigan
  - Columbia University Medical Center, New York, New York